CLINICAL TRIAL: NCT06263946
Title: Post Market Clinical Follow-up Study to Demonstrate the Efficacy, Safety, Acceptability and Quality of Life Implications of Essilor® Stellest® Spectacle Lenses in Slowing Myopia Progression in Children and Adolescents.
Brief Title: Essilor® Stellest® Lenses Multicentre European Study (SLOMES)
Acronym: SLOMES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS10337
Record Dates: First submitted 2024-01-29; First posted 2024-02-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: multicentre, European, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Essilor® Stellest® spectacle lenses (Other): patients will be asked to wear Essilor® Stellest® spectacle lenses for a full time wear (>12 hours daily) for 24 months
  Interventions: Device: Essilor® Stellest® spectacle lenses

INTERVENTIONS:
Device: Essilor® Stellest® spectacle lenses — patients will be asked to wear Essilor® Stellest® spectacle lenses more than 12 hours per day for 24 months.

SUMMARY:
The goal of this post-market clinical follow up Study is to demonstrate the efficacy, safety, acceptability, and quality of life implications of Essilor® Stellest® spectacle lenses in slowing myopia progression in European children and adolescents. Participants will receive Essilor® Stellest® at inclusion visit and will be asked for a full time wear (>12 hours daily) for 24 months. The primary endpoints are the change in axial length and cycloplegic autorefraction from baseline to 24 months compared to expected change based on axial length and refraction centile positions at baseline.

DETAILED DESCRIPTION:
The trial design is a multicentre, European, prospective, interventional study with single group assignment. The investigational medical device Essilor® Stellest® is a CE marked, myopia control spectacle lens. The trial period for all participants is 24 months. The recruiting period is 6 to 9 months depending on countries / sites for a total of 150 participants (50 in Ireland, 75 in France and 25 in The Netherlands).

The secondary objectives are:

* To evaluate the acceptability of Essilor® Stellest® spectacle lenses in slowing myopia progression.
* To evaluate the quality-of-life implications for children and adolescents.
* To evaluate the safety of Essilor® Stellest® spectacle lenses in slowing myopia progression.
* To evaluate the effect of Essilor® Stellest® spectacle lenses on choroidal thickness.

ELIGIBILITY:
Inclusion Criteria:

1. - Myopia as determined by cycloplegic autorefraction as follows:

   * Each meridian SER of plano to - 8;00 D in each eye
   * Astigmatism < 2.50 D
   * Anisometropia ≤ 1.50 D
2. - Monocular corrected VA of at least 0.2 LogMAR in both eyes
3. - Age: 6 - 16 years old, inclusive at the time of inclusion
4. - Ability to understand treatment and give valid assent
5. - Ability to comply with the protocol to get reliable study measurements

Exclusion Criteria:

1. - Concomitant or previous therapies for myopia
2. - Eye diseases/conditions:

   * Strabismus by cover test at near or distance
   * Any ocular disease that would influence refractive development e.g. retinal disease, cataract, ptosis
   * Any systemic or neurodevelopmental conditions that may influence refractive development
3. - Use of ocular or systemic medication which may affect myopia progression or visual acuity through known effects on retina, accommodation, or significant elevation of intraocular pressure
4. - Participation in another study which may influence vision or interfere with study assessments
5. - Myopia onset before 5 years of age
6. - Contact lens wearers

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2027-04-23 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in cycloplegic axial length | from baseline to 24 months
  in mm (millimeter) compared to expected change based on axial length at baseline (in each eye).
Change in cycloplegic autorefraction | from baseline to 24 months
  in D (Diopter) compared to expected change based on refraction centile positions at baseline (in each eye).

SECONDARY OUTCOMES:
Change in refraction progression centile | from 12 months to 24 months visits.
  compared to expected change based on refraction centile positions at baseline (in each eye).
Change in cycloplegic axial length | from baseline to 12 months and 24 months
  in mm (millimeter) compared to expected change based on axial length at baseline (in each eye).
Change in cycloplegic autorefraction | from baseline to 12 months and 24 months
  compared to expected change based on refraction centile positions at baseline (in each eye).
Change in refraction | during the first and second year of the Myopia Outcome Study of Atropine In Children (MOSAIC) study
  in D (Diopter) compared to that observed in control group participants of MOSAIC Study (myopia control trial conducted in Ireland from 2019 to 2023) (in each eye)
Change in axial length | during the first and second year (separate comparisons for each year) of the MOSAIC study.
  in mm (millimeter) compared to that observed in control group participants of the MOSAIC study (in each eye)
Change in choroidal thickness | during the first and second year (separate comparisons for each year) of the MOSAIC study.
  in μm (micrometre) compared to that observed in control group participants of the MOSAIC study (in each eye)
Change in refraction | during the first and second year (separate comparisons for each year) of the MOSAIC study.
  in D (Diopter) compared to children treated with 0.01% atropine in group participants of the MOSAIC study (in each eye)
Change in axial length vs atropine | during the first and second year (separate comparisons for each year) of the MOSAIC study.
  in mm (millimeter) compared to children treated with 0.01% atropine in group participants of the MOSAIC study (in each eye)
Change in choroidal thickness | during the first and second year (separate comparisons for each year) of the MOSAIC study
  in μm (micrometre) compared to children treated with 0.01% atropine in group participants of the MOSAIC study (in each eye)
Change in Paediatric Refractive Error Profile (PREP-2) score | from baseline (pre- Essilor® Stellest®) to 12 and 24 months (post- Essilor® Stellest®)
  Change in Paediatric Refractive Error Profile (PREP-2) score

CONTACTS AND LOCATIONS:
Overall Officials: Aude Couturier, Professor, Principal Investigator — Hôpital Fondation Adolphe de Rothschild - PARIS - FRANCE; Ian Flitcroft, Professor, Principal Investigator — Centre for Eye Research Ireland (CERI) - DUBLIN - IRELAND; Caroline Klaver, Professor, Principal Investigator — ERASMUS Medical Center - ROTTERDAM - NETHERLANDS
Locations (3):
- Hôpital Fondation Adolphe de Rothschild - Ophthalmology Department, Paris, France
- Centre for Eye Research Ireland (CERI) - TU DUBLIN, Dublin, Ireland
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039
- [Background] Bao J, Huang Y, Li X, Yang A, Zhou F, Wu J, Wang C, Li Y, Lim EW, Spiegel DP, Drobe B, Chen H. Spectacle Lenses With Aspherical Lenslets for Myopia Control vs Single-Vision Spectacle Lenses: A Randomized Clinical Trial. JAMA Ophthalmol. 2022 May 1;140(5):472-478. doi: 10.1001/jamaophthalmol.2022.0401. PMID 35357402
- [Background] Li X, Huang Y, Yin Z, Liu C, Zhang S, Yang A, Drobe B, Chen H, Bao J. Myopia Control Efficacy of Spectacle Lenses With Aspherical Lenslets: Results of a 3-Year Follow-Up Study. Am J Ophthalmol. 2023 Sep;253:160-168. doi: 10.1016/j.ajo.2023.03.030. Epub 2023 Apr 10. PMID 37040846